CLINICAL TRIAL: NCT01187992
Title: Full-dose Atorvastatin Versus Conventional Medical Therapy After Non-ST-elevation Acute Myocardial Infarction in Patients With Advanced Non-revascularisable Coronary Artery Disease
Brief Title: Full-dose Atorvastatin After Acute Coronary Syndrome (ACS) in Non-revascularisable Coronary Artery Disease
Acronym: APRIRE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Interim analysis showed significant effect in favour of full-dose atorvastatin.
Sponsor: San Filippo Neri General Hospital (Other)
Collaborators: Associazione Nazionale Medici Cardiologi Ospedalieri (Other)
Responsible Party: Prof. Furio Colivicchi, MD, FESC, Clinical Quality management Unit, Cardiovascular Department, San Filippo Neri Hospital, Rome Italy
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SFN/02/03/AL
Record Dates: First submitted 2010-08-24; First posted 2010-08-25 (Estimated); Last update posted 2010-08-25 (Estimated); Status verified 2010-05

CONDITIONS: Acute Coronary Syndrome; Coronary Artery Disease
Keywords: Atorvastatin; Acute coronary syndrome; Advanced coronary artery disease
MeSH Terms: conditions — Acute Coronary Syndrome; Coronary Artery Disease | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Full-dose atorovastatin (80 mg/d) (Experimental): For patients randomised to this arm, atorvastatin in the fixed dose of 80 mg/ day was started immediately after randomisation.
  Interventions: Drug: Atorvastatin
- Conventional medical treatment (No Intervention): For patients randomised to this arm, adherence to the National Cholesterol Education Program, Adult Treatment Panel III guidelines was required. In particular, in these patients,atorvastatin was started at the initial dosage of 20 mg/day immediately after randomisation. Subsequently, atorvastatin dosage was titrated in order to attain low-density lipoprotein cholesterol (LDL-C) levels <100 mg/dL (2.5 mmol/L).

INTERVENTIONS:
Drug: Atorvastatin — 80 mg/day
  Arms: Full-dose atorovastatin (80 mg/d)

SUMMARY:
This study was designed to test the hypothesis that the addition of full-dose atorvastatin (80 mg/day) to conventional medical treatment could reduce ischaemic recurrences after non-ST-elevation acute myocardial infarction (NSTE-AMI) in patients with severe and diffuse coronary artery disease (CAD) not amenable to any form of mechanical revascularisation.

ELIGIBILITY:
Inclusion Criteria:

* non-ST-segment elevation acute myocardial infarction.
* coronary angiography within 48 hours from admission.
* angiographic evidence of severe and diffuse coronary artery disease,not amenable to conventional direct revascularisation techniques by coronary artery bypass graft (CABG) or percutaneous coronary intervention (PCI).

Exclusion Criteria:

* ST-segment elevation acute myocardial infarction,
* clinical history of heart failure
* left ventricular ejection fraction <35%,
* any form of severe valvular dysfunction,
* previous implantation or indication to implant a cardioverter-defibrillator during the index admission,
* any increase in liver enzymes,
* history of any liver or muscle disease,
* renal failure with serum creatinine >2.5 mg/dL (221 mmol/L),
* need for continued use of intravenous medications to relieve anginal symptoms,
* presence of any major comorbidity with life expectancy <24 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2003-09; Primary Completion 2007-03 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiovascular events | 12 months
  The primary end point of the study was prospectively defined as the combination of cardiovascular death, non-fatal acute myocardial re-infarction (re-AMI) and disabling non-fatal stroke.

SECONDARY OUTCOMES:
Cardiovascular mortality | 12 months
Non-fatal acute myocardial re-infarction (re-AMI) | 12 months
Disabling non-fatal stroke | 12 months
New-onset heart failure | 12 months
Atrial fibrillation | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Furio Colivicchi, MD, Principal Investigator — Clinical Quality Mangement Unit, San Filippo Neri Hospital, Rome, Italy
Locations (1):
- San Filippo Neri General Hospital, Rome, Italy, Italy

REFERENCES:
- [Result] Colivicchi F, Tubaro M, Mocini D, Genovesi Ebert A, Strano S, Melina G, Uguccioni M, Santini M. Full-dose atorvastatin versus conventional medical therapy after non-ST-elevation acute myocardial infarction in patients with advanced non-revascularisable coronary artery disease. Curr Med Res Opin. 2010 Jun;26(6):1277-84. doi: 10.1185/03007991003751496. PMID 20367555